CLINICAL TRIAL: NCT01190644
Title: A Phase 2, Open-Label, Pharmacodynamic Study to Evaluate the Effect of Sotatercept (ACE-011) on Red Blood Cell Mass and Plasma Volume in Subjects With Solid Tumors
Brief Title: Study to Evaluate Effect of a Single Dose of Sotatercept (ACE-011) on Red Blood Cell Mass and Plasma Volume in Participants With Solid Tumors
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Isotope needed to conduct RBC/PV analysis (primary endpoint) no longer available from manufacturer. No alternatives available for use.
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 7962-016; ACE-011-ST-001 (Other: Celgene)
Record Dates: First submitted 2010-07-21; First posted 2010-08-27 (Estimated); Results first posted 2023-11-29 (Actual); Last update posted 2023-11-29 (Actual); Status verified 2023-11

CONDITIONS: Solid Tumors
Keywords: Red Blood Cell Mass; Plasma Volume; Solid Tumors
MeSH Terms: interventions — ACE-011

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Sotatercept (Experimental): Participants will receive a single 35 mg dose of sotatercept by subcutaneous (SC) injection on Day 1, Day 43, and Day 85.
  Interventions: Drug: Sotatercept

INTERVENTIONS:
Drug: Sotatercept — single 35 mg SC dose of sotatercept on study Day 1, Day 43, and Day 85
  Other Names: ACE 011

SUMMARY:
What hematopoietic precursor compartments as well as hemoglobin subtypes are affected by dosing with sotatercept (ACE-011)? Based upon a similar prior study with Procrit, Celgene has determined that all of these goals could be obtained by an intense 10-patient sotatercept (ACE-011) pharmacodynamic study, completed by two well-known experts in the red cell production field.

ELIGIBILITY:
Inclusion Criteria:

* Men and women ≥18 years of age.
* Histologically confirmed diagnosis of a solid tumor malignancy documented by cytology or biopsy.
* Presence of metastatic disease.
* Hemoglobin value between ≥8.0 to <11.0 g/dL (≥80 to <110 g/L).
* ≥28 days must have elapsed (prior to pre-dose red blood cell mass / plasma volume test) since previous treatment with erythropoiesis-stimulating agent (including concurrent treatment with intravenous [IV] iron).
* ≥28 days must have elapsed (prior to Day 1) since the last red blood cell transfusion and receipt of ≤2 units of blood in the past 56 days (prior to Day 1).
* Eastern Cooperative Oncology Group (ECOG) Performance status of 0 - 1.

Exclusion Criteria:

At the time of screening, participants who have any grade ≥3 toxicity (according to the currently active minor version of NCI CTCAE v4.0) except for the following disease-related toxicities:

* Hematological events - anemia, thrombocytopenia, neutropenia
* Non-hematological events - nausea, vomiting, fatigue, muscle or bone/joint pain

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2010-06-01 (Actual); Primary Completion 2012-09-18 (Actual); Study Completion 2012-10-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (3):
- United States (3):
  - Saint Agnes Healthcare, Baltimore, Maryland
  - Weinberg Cancer Institution at Franklin Square, Baltimore, Maryland
  - Pennsylvania Oncology, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Background] Cappellini MD, Porter J, Origa R, Forni GL, Voskaridou E, Galacteros F, Taher AT, Arlet JB, Ribeil JA, Garbowski M, Graziadei G, Brouzes C, Semeraro M, Laadem A, Miteva D, Zou J, Sung V, Zinger T, Attie KM, Hermine O. Sotatercept, a novel transforming growth factor beta ligand trap, improves anemia in beta-thalassemia: a phase II, open-label, dose-finding study. Haematologica. 2019 Mar;104(3):477-484. doi: 10.3324/haematol.2018.198887. Epub 2018 Oct 18. PMID 30337358
- See also: Merck Clinical Trials Information — http://www.merckclinicaltrials.com

RESULTS

PARTICIPANT FLOW:
Groups:
- Sotatercept: Participants received a single 35 mg dose of sotatercept by subcutaneous (SC) injection on Day 1, Day 43, and Day 85.
Period: Overall Study
Arm/Group | Sotatercept
Started | 5
Treated | 4
Completed | 2
Not Completed | 3
Not completed — Death | 2
Not completed — Disease progression | 1

BASELINE CHARACTERISTICS:
Arm/Group | Sotatercept
Number analyzed (Participants) | 5
Age, Continuous [Mean (Standard Deviation); unit: Years] | 63.8 (8.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 5
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 2
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Red Blood Cell Mass Following a Single Dose of Sotatercept
Description: Blood samples were to be collected at baseline (Day 1, pre-dose) and at one timepoint between Day 14 and Day 28, and isotope dilution techniques used, to measure the change from baseline in red blood cell mass following a single dose of sotatercept.
Time Frame: Baseline (Day 1, pre-dose) and one timepoint between Day 14 and Day 28
Population: No data were collected for Change from Baseline in Red Blood Cell Mass Following a Single Dose of Sotatercept.
Groups:
- Sotatercept: Participants received a single 35 mg dose of sotatercept by SC injection on Day 1, Day 43, and Day 85.
Arm/Group | Sotatercept
Number analyzed (Participants) | 0

2. Secondary Outcome: Change From Baseline in Plasma Volume Following a Single Dose of Sotatercept
Description: Blood samples were collected at baseline (Day 1, pre-dose) and at one timepoint between Day 14 and Day 28, and isotope dilution techniques used, to measure the change from baseline in plasma volume following a single dose of sotatercept.
Time Frame: Baseline (Day 1, pre-dose) and one timepoint between Day 14 and Day 28
Population: All participants who received at least one dose of study treatment and had data for Change from Baseline in Plasma Volume Following a Single Dose of Sotatercept
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | Sotatercept
Number analyzed (Participants) | 2
mL | -239.50 (219.91)

3. Secondary Outcome: Change From Baseline in Absolute Reticulocyte Count
Description: Blood samples were to be collected at baseline (Day 1, pre-dose) and at Day 211 to measure the change from baseline in absolute reticulocyte count.
Time Frame: Baseline (Day 1, pre-dose) and Day 211
Population: No data were collected for Change from Baseline in Absolute Reticulocyte Count.
Arm/Group | Sotatercept
Number analyzed (Participants) | 0

4. Secondary Outcome: Change From Baseline in Erythropoietin Levels
Description: Blood samples were collected at baseline (Day 1, pre-dose) and at Day 211 to measure the change from baseline in erythropoietin levels.
Time Frame: Baseline (Day 1, pre-dose) and Day 211
Population: All participants who received at least one dose of study treatment and had data for Change from Baseline in Erythropoietin Levels
Measure: Mean (Full Range); unit: IU/L
Arm/Group | Sotatercept
Number analyzed (Participants) | 1
IU/L | 11.30 [11.3 to 11.3]

5. Secondary Outcome: Change From Baseline in Hemoglobin Subtype A Following a Single Dose of Sotatercept
Description: Blood samples were collected at baseline (Day 1, pre-dose) and on Day 29, and hemoglobin electrophoresis used, to measure the change from baseline in hemoglobin subtype A following a single dose of sotatercept.
Time Frame: Baseline (Day 1, pre-dose) and Day 29
Population: All participants who received at least one dose of study treatment and had data for Change from Baseline in Hemoglobin Subtype A Following a Single Dose of Sotatercept
Measure: Mean (Full Range); unit: Percentage of hemoglobin subtype A
Arm/Group | Sotatercept
Number analyzed (Participants) | 1
Percentage of hemoglobin subtype A | 0.0 [0.0 to 0.0]

6. Secondary Outcome: Change From Baseline in Hemoglobin Subtype A2 Following a Single Dose of Sotatercept
Description: Blood samples were collected at baseline (Day 1, pre-dose) and on Day 29, and hemoglobin electrophoresis used, to measure the change from baseline in hemoglobin subtype A2 following a single dose of sotatercept.
Time Frame: Baseline (Day 1, pre-dose) and Day 29
Population: All participants who received at least one dose of study treatment and had data for Change from Baseline in Hemoglobin Subtype A2 Following a Single Dose of Sotatercept
Measure: Mean (Full Range); unit: Percentage of hemoglobin subtype A2
Arm/Group | Sotatercept
Number analyzed (Participants) | 1
Percentage of hemoglobin subtype A2 | 0.0 [0.0 to 0.0]

7. Secondary Outcome: Change From Baseline in Hemoglobin Subtype C Following a Single Dose of Sotatercept
Description: Blood samples were collected at baseline (Day 1, pre-dose) and on Day 29, and hemoglobin electrophoresis used, to measure the change from baseline in hemoglobin subtype C following a single dose of sotatercept.
Time Frame: Baseline (Day 1, pre-dose) and Day 29
Population: All participants who received at least one dose of study treatment and had data for Change from Baseline in Hemoglobin Subtype C Following a Single Dose of Sotatercept
Measure: Mean (Full Range); unit: Percentage of hemoglobin subtype C
Arm/Group | Sotatercept
Number analyzed (Participants) | 1
Percentage of hemoglobin subtype C | 0.0 [0.0 to 0.0]

8. Secondary Outcome: Number of Participants Who Experienced One or More Adverse Events (AEs)
Description: An AE is any untoward medical occurrence in a study participant administered a pharmaceutical product that does not necessarily have to have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign, symptom, or disease temporally associated with the use of a medicinal product, whether or not related to the medicinal product.
Time Frame: Up to approximately 7 months
Population: All participants who received at least one dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Sotatercept
Number analyzed (Participants) | 4
Participants | 4

ADVERSE EVENTS:
Time Frame: Up to approximately 7 months
Description: The safety analysis population included all participants who received at least one dose of study treatment. The analysis population for All-Cause Mortality included all enrolled participants.
Groups:
- Sotatercept 35 mg: Participants received a single 35 mg dose of sotatercept by SC injection on Day 1, Day 43, and Day 85.
Arm/Group | Sotatercept 35 mg
All-Cause Mortality (participants affected / at risk) | 2/5
Serious Adverse Events (participants affected / at risk) | 3/4
Other Adverse Events (participants affected / at risk) | 4/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sotatercept 35 mg (N=4)
CARDIO-RESPIRATORY ARREST (Cardiac disorders) | 1 (1)
CARDIOGENIC SHOCK (Cardiac disorders) | 1 (1)
ABDOMINAL PAIN (Gastrointestinal disorders) | 1 (2)
PNEUMOPERITONEUM (Gastrointestinal disorders) | 1 (1)
DEVICE DISLOCATION (General disorders) | 1 (1)
INFECTED SKIN ULCER (Infections and infestations) | 1 (1)
PROCEDURAL PAIN (Injury, poisoning and procedural complications) | 1 (2)
DEHYDRATION (Metabolism and nutrition disorders) | 1 (1)
HYPONATRAEMIA (Metabolism and nutrition disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sotatercept 35 mg (N=4)
ANAEMIA (Blood and lymphatic system disorders) | 1 (1)
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 1 (1)
MYOCARDIAL INFARCTION (Cardiac disorders) | 1 (1)
ABDOMINAL DISTENSION (Gastrointestinal disorders) | 1 (1)
ASCITES (Gastrointestinal disorders) | 1 (1)
CONSTIPATION (Gastrointestinal disorders) | 1 (2)
GASTROOESOPHAGEAL REFLUX DISEASE (Gastrointestinal disorders) | 1 (1)
NAUSEA (Gastrointestinal disorders) | 1 (1)
VOMITING (Gastrointestinal disorders) | 3 (3)
OEDEMA PERIPHERAL (General disorders) | 2 (2)
DEVICE RELATED INFECTION (Infections and infestations) | 1 (1)
ESCHERICHIA INFECTION (Infections and infestations) | 1 (1)
NASOPHARYNGITIS (Infections and infestations) | 1 (1)
ORAL CANDIDIASIS (Infections and infestations) | 1 (1)
WOUND INFECTION STAPHYLOCOCCAL (Infections and infestations) | 1 (1)
PROCEDURAL PAIN (Injury, poisoning and procedural complications) | 1 (1)
DEHYDRATION (Metabolism and nutrition disorders) | 1 (1)
HYPERGLYCAEMIA (Metabolism and nutrition disorders) | 1 (1)
HYPOCALCAEMIA (Metabolism and nutrition disorders) | 1 (2)
HYPOKALAEMIA (Metabolism and nutrition disorders) | 1 (1)
HYPOMAGNESAEMIA (Metabolism and nutrition disorders) | 1 (2)
MUSCULOSKELETAL PAIN (Musculoskeletal and connective tissue disorders) | 1 (1)
HEADACHE (Nervous system disorders) | 1 (1)
ANXIETY (Psychiatric disorders) | 1 (1)
INSOMNIA (Psychiatric disorders) | 1 (1)
DYSPNOEA EXERTIONAL (Respiratory, thoracic and mediastinal disorders) | 1 (1)
ERYTHEMA (Skin and subcutaneous tissue disorders) | 1 (1)
SKIN ULCER (Skin and subcutaneous tissue disorders) | 1 (1)
HYPERTENSION (Vascular disorders) | 1 (1)
HYPOTENSION (Vascular disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor will comply with the requirements for publication of study results. In accordance with standard editorial and ethical practice, the sponsor will generally support publication.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2012-03-05): https://cdn.clinicaltrials.gov/large-docs/44/NCT01190644/Prot_SAP_000.pdf